CLINICAL TRIAL: NCT03996005
Title: Evaluation of an Alternative Treatment of Localized Prostate Cancer by Guided MRI Transurtral Ultrasound With 1-year Control of the Absence of Cancer
Brief Title: MRI- Guided Transurethral Ultrasound Ablation of Localized Prostate Cancer
Acronym: MRI-TULSAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7429
Record Dates: First submitted 2019-06-19; First posted 2019-06-24 (Actual); Results first posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: MRI Guided Transurethral Ultrasound Ablation; Localized Prostate Cancer; Ablation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRI Guided Transurethral Ultrasound (Experimental): Magnetic Resonance Imaging-Guided Transurethral Ultrasound Ablation of Prostate Tissue
  Interventions: Procedure: Magnetic Resonance Imaging-Guided Transurethral Ultrasound Ablation of Prostate Tissue

INTERVENTIONS:
Procedure: Magnetic Resonance Imaging-Guided Transurethral Ultrasound Ablation of Prostate Tissue — Magnetic Resonance Imaging-Guided Transurethral Ultrasound Ablation of Prostate Tissue

SUMMARY:
Primary purpose :

Evaluation of the efficiency and safety of an alternative global prostate treatment in localized prostate cancer.

Primary Objective:

Absence of clinically significant cancer (CSC) on control biopsy at 1-year follow-up.

Secondary Objectives:

1. Biochemical response
2. Presence of any CSC on biopsy at 1- and 2-year follow-up
3. Radical treatment free survival
4. Adverse events, clinical tolerance
5. Urinary continence
6. Erectile function
7. Quality of life

ELIGIBILITY:
Inclusion Criteria:

* Male patient ≥ 50 years old
* Histologically confirmed adenocarcinoma of the prostate
* Gleason ≤ 7 (3 + 4) ; Grade group ≤ 2 according to Epstein
* Clinically <T3, N0, M0
* PSA < 15 ng/mL
* Prostate volume <100g
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Life expectancy higher than 12 months in the judgement of the investigator
* Radiological TNM (prostate MRI) T ≤ 2 (absence of extra-capsular extension, absence of seminal vesicle invasion), N = 0, M = 0
* First line of treatment or relapse after initial radiotherapy
* Willing to give signed, informed consent freely
* Able to adhere to the follow-up schedule and other protocol requirements.

Exclusion Criteria:

* Contraindication to MRI
* Contraindication to general anesthesia
* Presence or history of any other malignancy except for non-melanoma skin cancer adequately treated at least 2 years before study entry
* Unreversible haemostasis disorder

Min Age: 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thibault TRICARD, MD, Principal Investigator — University Hospital, Strasbourg, France
Locations (1):
- Hôpitaux Universitaires de strasbourg, Strasbourg, France

REFERENCES:
- [Result] Tricard T, Cazzato RL, Schroeder A, De Mathelin M, Barhoumi C, Gaillard V, Sauleau E, Gangi A, Lang H. Magnetic Resonance Imaging-guided Transurethral Ultrasound Ablation (TULSA) of Localized Prostate Cancer: A prospective Trial. J Vasc Interv Radiol. 2025 Sep;36(9):1401-1408. doi: 10.1016/j.jvir.2025.05.024. Epub 2025 May 27. PMID 40441432

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MRI Guided Transurethral Ultrasound
Started | 25
Completed | 24
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | MRI Guided Transurethral Ultrasound
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.8 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 24
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Clinically significant cancer (CSC) on biopsy [Count of Participants; unit: Participants] — Population: 1 patient was deemed unfit for biopsy
  Participants
    number analyzed (Participants) | 23
    (all) | 10

OUTCOME MEASURES:

1. Primary Outcome: Absence of Clinically Significant Cancer (CSC) on Control Biopsy at 1-year Follow-up.
Description: Clinically significant cancer (CSC) defined by at least one of the following criteria:
  * Gleason score ≥ 7
  * cancer core length > 3 mm regardless of Gleason score
  * > 2 positive cores.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | MRI Guided Transurethral Ultrasound
Number analyzed (Participants) | 23
Participants | 8

ADVERSE EVENTS:
Time Frame: 1 year
Description: old study, no possibility of MedDRA coding for non-serious AE
Arm/Group | MRI Guided Transurethral Ultrasound
All-Cause Mortality (participants affected / at risk) | 1/25
Serious Adverse Events (participants affected / at risk) | 3/25
Other Adverse Events (participants affected / at risk) | 0/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MRI Guided Transurethral Ultrasound (N=25)
renal failure (Renal and urinary disorders) | 1
urinary retention (Renal and urinary disorders) | 1
Coronary artery disease (Cardiac disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-20): https://cdn.clinicaltrials.gov/large-docs/05/NCT03996005/Prot_SAP_000.pdf